CLINICAL TRIAL: NCT03732456
Title: Predictors of Post-operative Pain in Shoulder Surgery, a Prospective Observational Study
Brief Title: Post-operative Pain After Shoulder Surgery
Status: Completed | Type: Observational
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Marie Awad, Professor of Anesthesiology, Interim Chairperson, American University of Beirut Medical Center
Other Study IDs: BIO-2018-0083
Record Dates: First submitted 2018-11-02; First posted 2018-11-06 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Pain, Shoulder
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Shoulder surgery and post-op pharmacological treatment — Usual care surgery (shoulder arthroscopy) and post-operative pain management protocol

SUMMARY:
A prospective observational study conducted at the American University of Beirut Medical center that targets patients undergoing shoulder surgeries. It is conducted to to prospectively collect patient, surgery and anesthesia-related variables and perform correlation studies with postoperative pain severity, patients' satisfaction and analgesic consumption following shoulder surgery.

In addition, identifying predictors for postoperative pain will contribute to adjust pain management protocols as per surgical and patients' factors.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients > 18 years old admitted to the American University of Beirut - Medical Center for any shoulder surgery

Exclusion Criteria:

* Patients suffering of opioids addiction (or previous history of addiction) or drug abuse.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients older than 18 years of age and admitted to the American University of Beirut Medical Center for any shoulder surgery
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Postoperative change in pain intensity (NRS pain scale) | 24 hours, 3 days and one week after surgery
  Asses the change in pain intensity after the surgery using the NRS pain score (0-10)
Postoperative change in satisfaction with pain management (NRS satisfaction scale) | 24 hours, 3 days and one week after surgery
  Asses the change in satisfaction with the pain management protocol using the NRS satisfaction score (0-10)
Postoperative analgesic consumption | Over one week
  Analgesic consumption over one week after the surgery
Postoperative functional level (QuickDASH questionnaire) | One week after surgery
  The QuickDASH questionnaire includes questions about the symptoms and ability to do certain activities

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon